CLINICAL TRIAL: NCT01560962
Title: Efficacy of Over the Counter (OTC) Povidone-Ioldine 5% for Treatment of Acute or Chronic Blepharitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: research staffs unable to continue.
Sponsor: Southern California Institute for Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: blepharitis
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Blepharitis
MeSH Terms: conditions — Blepharitis | interventions — Povidone-Iodine; Azithromycin

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- PI vs no intervention (Other): In group one, 25 patients will be instructed to scrub the lid margin of one eye with 5% PI twice daily for 10 days and the other eye with no intervention.
  Interventions: Drug: povidone iodine; Other: No Intervention
- PI vs hygiene (Other): In group two, 25 patients will be instructed to scrub the lid margin of one eye with 5% PI and the other eye will receive warm soaked eyelid wash.
  Interventions: Drug: povidone iodine; Other: warm soaked eyelid wash
- PI vs azasite (Other): In group three, 25 patients will be instructed to scrub the lid margin of one eye with 5% PI and the other eye will receive 1 drop of azithromycin ophthalmic solution twice daily for 10 days.
  Interventions: Drug: povidone iodine; Drug: Azithromycin
- PI vs tobradex (Other): In group four, 25 patients will be instructed to scrub the lid margin of one eye with 5% PI and the other eye will receive tobradex ointment applied to the lid margin.
  Interventions: Drug: povidone iodine; Drug: tobramycin-dexmethasone

INTERVENTIONS:
Drug: povidone iodine — over the counter (OTC) 5% povidone iodine (PI)
Other: No Intervention
  Arms: PI vs no intervention
Drug: Azithromycin
  Other Names: Azasite
  Arms: PI vs azasite
Drug: tobramycin-dexmethasone
  Arms: PI vs tobradex
Other: warm soaked eyelid wash
  Arms: PI vs hygiene

SUMMARY:
Objective: To determine the preliminary outcome of external over the counter (OTC) povidone iodine (PI) application in the management of chronic and acute blepharitis vs. currently clinically accepted medical regimen, i.e. eyelid hygiene, antibiotic drops, or antibiotic/steroid ointments.

Methodology: One hundred adult patients with chronic and acute blepharitis will be enrolled and randomized into four groups.

In group one, 25 patients will be instructed to scrub the lid margin of one eye with 5% PI twice daily for 10 days and the other eye with no intervention.

In group two, 25 patients will be instructed to scrub the lid margin of one eye with 5% PI and the other eye will receive warm soaked eyelid wash.

In group three, 25 patients will be instructed to scrub the lid margin of one eye with 5% PI and the other eye will receive 1 drop of azithromycin ophthalmic solution twice daily for 10 days.

In group four, 25 patients will be instructed to scrub the lid margin of one eye with 5% PI and the other eye will receive tobradex ointment applied to the lid margin.

Subjective variables assessed included itchiness, foreign body sensation and eyelid edema (grade 0-4). Objective variables assessed included lid margin redness, meibomian gland plugging and presence/absence of collarets (grade 0-4). Cultures of lid margin at the initiation and at the cessation of treatment were obtained.

DETAILED DESCRIPTION:
Final statiscial analysis for subjective and objective numerical values following treatment for each group of subjects (group 2,3,4) should show equal or almost equal efficacy in treatment of blepharitis.

ELIGIBILITY:
Inclusion Criteria:

* All potential subjects with symptomatic blepharitis examined to have blepharitis with healthy mental status, able to give consent, with/without co-existing medical consitions will be considered.

Exclusion Criteria:

* All subjects with history and/or probable history of allergic reaction to povidine-iodine, azithromycin, & tobramycin/dexamethasone and all subjects who have mental disability and are unable to give direct consent will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
meibomian gland plugging | 01/12 to 01/13
  Variables of interest will include:
  A. Subjective Measures including patient-rated symptom scores for 1. Itching (grade 0-3) 2. foreign body sensation (grade 0-3) 3. ocular dryness (grade 0-3) 4. ocular burning (grade 0-3) and 5. swollen eyelids (grade 0-3) B. Objective Measures: Evaluation of 1. lid margin redness (grade 0-3) 2. meibomian gland plugging (grade 0-3) and 3. Presence of collarets and scurfs (Grade 0-3) 4. Cultures of eyelid margin at the start and at the conclusion of treatment at 10 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Veterans Affairs Long Beach Healthcare System, Long Beach, California, United States